CLINICAL TRIAL: NCT01340716
Title: Effects of Tai Chi Chuan on Blood Pressure, Respiratory Muscle Strength and Functional Capacity in Patients After Recent Acute Myocardial Infarction: a Randomized Clinical Trial
Brief Title: Effects of Tai Chi Chuan in Patients After Recent Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GPPG 100531
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2016-02

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stretching exercise (Active Comparator): patients in this group held three weekly classes of 60 minutes during 12 weeks of Tai Chi Chuan, Yang style.
  Interventions: Other: stretching exercise
- Tai Chi Chuan exercise (Experimental): patients in this group held weekly classes of two stretching for 12 weeks.
  Interventions: Other: Tai Chi Chuan exercise

INTERVENTIONS:
Other: Tai Chi Chuan exercise — patients in this group held three weekly classes of 60 minutes during 12 weeks of Tai Chi Chuan, Yang style. The exercises will be mild to moderate (HR 60 to 75% of HR Max). Slow movements combined with exercises and maintained using your own body weight.
  Arms: Tai Chi Chuan exercise
Other: stretching exercise — patients in this group held weekly classes of two stretching for 12 weeks.
  Arms: stretching exercise

SUMMARY:
This is a randomized Clinical Trial to assess the effects of Tai Chi Chuan on blood pressure, respiratory muscle strength and functional capacity in patients after recent acute myocardial infarction.

DETAILED DESCRIPTION:
Background:Patients with a recent myocardial infarction (MI) present a reduction in functional capacity expressed as a decrease in peak oxygen consumption (VO2 peak). The impact of a Tai Chi Chuan (TCC) cardiac rehabilitation program for patients recovering from recent MI has yet to be assessed. Our goal is to evaluate functional capacity after a TCC-based cardiac rehabilitation program in patients with recent MI.

Methods: A single-blind randomized clinical trial was conducted. The researchers who performed the tests were blinded to group allocation. Between the 14th and 21st days after hospital discharge, all patients performed a cardiopulmonary exercise testing and a laboratory blood workup. Mean age was similar (56 ± 9 years in the TCC group and 60 ± 9 years in the control group). Patients allocated to the intervention group performed 3 weekly sessions of TCC Beijin style for 12 weeks (n = 31). The control group participated in 3 weekly sessions of full-body stretching exercises (n = 30).

ELIGIBILITY:
Inclusion Criteria:

* Recent acute myocardial infarction
* Age 45 and 75 years.
* admission until 20 days after hospital discharge
* With physical conditions for a cardiac rehabilitation program with exercise.

Exclusion Criteria:

* Unstable angina
* Severe congestive heart failure
* Severe lung disease
* Altered response of blood pressure to stress

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
functional capacity | Change from Baseline in functional capacity at 90 days
  cardiopulmonary exercise testing (VO2)

SECONDARY OUTCOMES:
respiratory muscle strength | Change from Baseline in respiratory muscle strength at 90 days
  PImax e PEmax were obtained using a pressure tansducer
Ambulatory blood pressure in 24 hours | Change from Baseline in blood pressure at 90 days
  24-hour blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Rosane Nery, Principal Investigator — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nery RM, Zanini M, de Lima JB, Buhler RP, da Silveira AD, Stein R. Tai Chi Chuan improves functional capacity after myocardial infarction: A randomized clinical trial. Am Heart J. 2015 Jun;169(6):854-60. doi: 10.1016/j.ahj.2015.01.017. Epub 2015 Mar 13. PMID 26027624